CLINICAL TRIAL: NCT01186471
Title: A Double-Blind, Placebo-Controlled, Randomized Three-Way Crossover Study to Investigate The Effect of Nicotine on Arousal, Standard Cognitive Tasks And Social Cognition in Patients With Schizophrenia (Smoking and Non-Smoking)
Brief Title: The Effect of Nicotine on Arousal, Cognition and Social Cognition in Schizophrenic Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Clinical Scientist/Director, Experimental Medicine, Janssen Pharmaceutica N.V., Belgium
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: CR017263
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia; Cognition Disorders
Keywords: Symptomatic treatment; Cognition; Cognitive deficits; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 001 (Experimental): A643 (nicotine) 1mg oromucosal nicotine spray- three times daily during each treatment period
  Interventions: Other: A643 (nicotine)
- 002 (Experimental): A643 (nicotine) 2mg oromucosal nicotine spray- three times daily during each treatment period
  Interventions: Other: A643 (nicotine)
- 003 (Placebo Comparator): placebo placebo - three times daily during each treatment period
  Interventions: Drug: placebo

INTERVENTIONS:
Other: A643 (nicotine) — 1mg oromucosal nicotine spray- three times daily during each treatment period
  Arms: 001
Other: A643 (nicotine) — 2mg oromucosal nicotine spray- three times daily during each treatment period
  Arms: 002
Drug: placebo — placebo - three times daily during each treatment period
  Arms: 003

SUMMARY:
This study in patients with stable schizophrenia will investigate the effect of nicotine on arousal, cognitive task and social cognition after acute dose administration.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor patient knows the name of the assigned drug), placebo-controlled, randomized (study drug assigned by chance), three-way-crossover trial (patients may receive different interventions sequentially during the trial) in patients with stable schizophrenia. The three-way-crossover treatment phase will consist of three blinded treatment periods separated by a wash out period (the period allowed for the entire administered drug to be eliminated from the body) of 2 to 7 days. The study duration for each patient will be approximately 8 weeks. Each patient enrolled will be randomized to receive Treatment A (1mg nicotine per dosing), Treatment B (2mg nicotine per dosing) or Treatment C (placebo) during one of their treatment period. The study drug (nicotine or placebo) will be administered three times daily on Day 1 of each treatment phase as a mouth spray, separated 2 to 3 hours from each other (i.e. 0h; and 2 to 3h; and 4 to 6h post first dosing). Three different blocks of cognitive assessments will follow, one after each drug administration. Safety evaluations include adverse event monitoring, vital signs and clinical laboratory tests. Each patient participating will receive 3 identical study drug administrations per dosing day (2 to 3 hours from each other), resulting in an overall dose of 3 mg nicotine (Treatment A), 6 mg nicotine (Treatment B) or 0 mg nicotine (Treatment C) per dosing day. By the end of the study, after the 3-way crossover, each patient will have received 9 mg nicotine via mouth spray.

ELIGIBILITY:
Inclusion Criteria:

* In- or outpatients with schizophrenia stably treated (same primary medication) for at least 2 months with antipsychotic therapy (treatment with more than 1 antipsychotic drug is acceptable provided dose levels have been stable for > 2 months). Fluctuations in dose levels of the primary antipsychotic treatment are acceptable provided the dose levels remain constant as from 2 weeks prior to dosing
* A known (by the site) disease history of at least 12 months
* DSM-IV criteria for Schizophrenia
* Willing to be hospitalized during the treatment periods of the study
* Body mass index (BMI) between 18 and 35 kg/m2, inclusive (BMI = weight/height2)
* Women must be: postmenopausal (for at least 12 months), surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), abstinent (at the discretion of the investigator/per local regulations), or if sexually active, be practicing a highly effective method of birth control and must agree to continue to use the same method of contraception throughout the study
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at admission (each study period)
* Smoking on average a minimum of 15 cigarettes (or equivalent) per day within 6 months prior to study drug administration (only for Cohort 1)

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding
* Clinically significant abnormal values for clinical chemistry, hematology or urinalysis at screening. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to the investigator, are acceptable. Values of alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2 fold ULN will be allowed
* Clinically significant abnormal physical examination, vital signs or 12-lead ECG at screening
* A DSM-IV axis I diagnosis other than schizophrenia that has been the focus of treatment or cause of disability in the last 6 months (such as Major Depressive Episode)
* Evidence of substance dependence other than nicotine (DSM-IV) in the last 6 months
* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, unmanaged high BP, hematological disease, bronchospastic respiratory disease, renal or hepatic insufficiency, Parkinson's disease, infection (HIV, Hepatitis C), or any other illness that the Investigator considers should exclude the subject (Subjects with mild hypertension, lipid abnormalities, diabetes mellitus or thyroid disease are allowed if no significant treatment changes were required in the past 6 months)
* Use of anti-parkinsonian agents in the past 2 months
* Suicidal risk (assessed by the investigator), prior attempts to suicide, command hallucinations and / or hopelessness
* Smoking cigarettes (or equivalents) or the use of nicotine based products within 3 months prior to study drug administration (only for Cohort 2)
* Current use of any medication for smoking cessation such as nicotine replacement therapy, bupropion or varenicline
* History of epilepsy or fits or unexplained black-outs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-05; Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Event related potentials (P50, P300, N100) and measures of standard cognition and social cognition | 1 hour post dose

SECONDARY OUTCOMES:
Nicotine exposure | predose and 5 min post each dosing

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.